CLINICAL TRIAL: NCT02379195
Title: T Cell Therapy in Combination With Peginterferon for Patients With Metastatic Melanoma
Brief Title: Peginterferon and TIL Therapy for Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Prof., MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM1413
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; aldesleukin; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): All patients receive the same treatment.
  All patients are hospitalized during treatment (approximately 3 weeks) and receive treatment only once.
  The patients are admitted to hospital day -8 and receive lymphodepleting chemotherapy (cyclophosphamide and fludarabine) on day -7 to day -1.
  The TILs are infused on day 0 and Interleukin-2 therapy are administered on day 0 to day 5.
  Interleukin-2 are administered in an i.v. continuous decrescendo regimen starting approximately 6 hours after TIL infusion with a duration of approximately 5 days
  Subcutaneous injections of peginterferon alpha 2b are administered three time (day -2, day 7 and day 14)
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: TIL infusion; Drug: Interleukin-2; Drug: Peginterferon alfa-2b

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg are administered i.v on day -7 and -6
Drug: Fludarabine — Fludarabine 25 mg/m2 are administered i.v on day -5 to -1
  Other Names: Fludarabinephosphate; Fludara
Biological: TIL infusion — The maximum number of expanded TILs are infused over 30-45 min on day 0
  Other Names: T cell infusion
Drug: Interleukin-2 — Interleukin-2 are administered as a continuous i.v. infusion in a decrescendo regimen (18 MIU/m2 IL-2 over 6 hours, 18 MIU/m2 IL-2 over 12 hours, 18 MIU IL-2 over 24 hours followed by 4.5 MIU/m2 IL-2 over another 24 hours for three days)
  Other Names: IL-2; Proleukin
Drug: Peginterferon alfa-2b — Peginterferon alpha-2b, 3 microgram/kg are administered as subcutaneous injection on day -2, day 7 and day 14.
  Other Names: PegIntron

SUMMARY:
Adoptive T cell therapy with tumor infiltrating lymphocytes (TIL) has achieved impressive clinical results with durable complete responses in patients with metastatic melanoma. The TILs are isolated from the patients own tumor tissue followed by in vitro expansion and activation for around 4-6 weeks. Before TIL infusion the patients receive 1 week of preconditioning chemotherapy with cyclophosphamide and fludarabine. After TIL infusion Interleukin-2 are administered to support T cell activation and proliferation in vivo.

In this trial the therapy is combined with peginterferon (the pegylated form of interferon alpha 2b). Interferon alpha has immunomodulatory effects and is known to upregulate HLA expression on melanoma cells and are hypothesized to synergize with TIL therapy.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed unresectable stage III or stage IV metastatic melanoma Metastasis available for surgical resection (about 2 cm3) and residual measurable disease after resection

ECOG performance status 0-1

Life expectancy ≥ 3 months

No significant toxicity from prior treatments

Adequate renal, hepatic and hematologic function

Women of childbearing potential (WOCBP) and men in a sexual relationship with a WOCBP must be using an effective method of contraception during treatment and for at least 6 months after completion af treatment.

Able to comprehend the information given and willing to sign informed consent

-

Exclusion Criteria:

Other Malignancies, unless followed for ≥ 5 years with no sign of disease, except squamous cell carcinoma or adequately treated carcinoma in situ colli uteri.

Cerebral metastasis. Patients with previously treated CNS metastases can participate if CNS metastases are surgically removed or treated with stereotactic radiosurgery and stable ≥ 28 days after treatment measured by MRI. Patients with asymptomatic, stable and untreated CNS metastasis can in be included according to investigators and sponsors decision.

Patients with ocular melanoma

Severe allergies, history of anaphylaxis or known allergies to the administered drugs.

Serious medical or psychiatric comorbidity

Creatinine clearance < 70 ml/min

Acute or chronic infection with e.g. HIV, hepatitis, tuberculosis

Severe and active autoimmune disease

Pregnant and nursing women

Need for immunosuppressive treatment, e.g. corticosteroids or methotrexate

Concomitant treatment with other experimental drugs

Patients with uncontrolled hypercalcemia

Less than four weeks since prior systemic antineoplastic treatment at the time of treatment.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Prof, PhD, MD, Study Director — Center for Cancer Immune Therapy, Dept of Hematology/Oncology, Copenhagen University Hospital Herlev, Herlev Ringvej 75, DK-2730 Herlev, Denmark; Rikke Andersen, MD, Principal Investigator — Center for Cancer Immune Therapy, Dept of Hematology/Oncology, Copenhagen University Hospital Herlev, Herlev Ringvej 75, DK-2730 Herlev, Denmark
Locations (1):
- Center for Cancer Immune Therapy, Dept. of Haematology/Oncology, Copenhagen, Herlev, Denmark

REFERENCES:
- [Derived] Borch TH, Andersen R, Ellebaek E, Met O, Donia M, Svane IM. Future role for adoptive T-cell therapy in checkpoint inhibitor-resistant metastatic melanoma. J Immunother Cancer. 2020 Jul;8(2):e000668. doi: 10.1136/jitc-2020-000668. PMID 32747469

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited from Danish melanoma centers.
Groups:
- Arm A: TIL + IFNalpha: The patients are admitted to hospital day -8 and receive lymphodepleting chemotherapy with cyclophosphamide 60 mg/kg on day -7 and -6 and fludarabine 25 mg/m2 on day -5 to day -1.
  TIL infusion: The maximum number of expanded TILs are infused over 30-45 min on day 0
  Interleukin-2: Interleukin-2 are administered as a continuous i.v. infusion in a decrescendo regimen (18 MIU/m2 IL-2 over 6 hours, 18 MIU/m2 IL-2 over 12 hours, 18 MIU IL-2 over 24 hours followed by 4.5 MIU/m2 IL-2 over another 24 hours for three days)
  Peginterferon alfa-2b: Peginterferon alpha-2b, 3 microgram/kg are administered as subcutaneous injection on day -2, day 7 and day 14.
Period: Overall Study
Arm/Group | Arm A: TIL + IFNalpha
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm A: TIL + IFNalpha
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 57 [42 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events/Serious Adverse Events
Description: Determine the safety of the administration of peginterferon in combination with TIL therapy including lymphodepleting chemotherapy and Interleukin-2 by reporting adverse events according to CTCAE v. 4.0
Time Frame: 0-24 weeks
Population: 12 patients were treated with TIL.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: TIL + IFNalpha
Number analyzed (Participants) | 12
Participants
  Adverse events | 12
  Treatment-related adverse events | 12
  Serious adverse events | 4

2. Secondary Outcome: Treatment Related Immune Responses
Description: Number of participants with detectable in vitro immune responses in the TIL infusion product using intracellular flow cytometry.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: TIL + IFNalpha
Number analyzed (Participants) | 12
Participants | 6

3. Secondary Outcome: Objective Response Rate
Description: Clinical responses will be evaluated by RECIST 1.1 (Response Criteria In Solid Tumors Criteria version 1.1) and assessed by CT scan. Complete response (CR), disapperance of all lesions; Partial response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective response (OR) = CR + PR
Time Frame: Up to 36 months
Population: 12 patients were treated with TIL. 1 patient was not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: TIL + IFNalpha
Number analyzed (Participants) | 11
Participants | 2

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS), defined as time from treatment initiation to death, described using the Kaplan Meier method
Time Frame: Up to 36 months
Population: 12 patients were treated with TIL. 1 patient was not evaluable.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: TIL + IFNalpha
Number analyzed (Participants) | 11
months | 11.75 [0.13 to 27.33]

5. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS), defined as the time from treatment initiation to disease progression, relapse or death due to any cause, which ever comes first, will be described with the Kaplan Meier method.
Time Frame: Up to 36 months
Population: 12 patients were treated with TIL. 1 patient was not evaluable.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: TIL + IFNalpha
Number analyzed (Participants) | 11
months | 2.8 [0.13 to 18.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from starting treatment until 24 weeks after TIL infusion.
Description: Adverse events were recorded in open-ended discussion and through scoring of adverse events according to AE recording forms by the treating physician.
Arm/Group | Arm A: TIL + IFNalpha
All-Cause Mortality (participants affected / at risk) | 8/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: TIL + IFNalpha (N=12)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1) — Oral/eosophagitis due to candidiasis
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1) — After restitution, patient had a period of low platelet count, decreased leukocytes and anemia. Spontaneously normalized.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm A: TIL + IFNalpha (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (12)
Infection (Infections and infestations) | 7 (7) — Verified infections
Fatique (General disorders) | 12 (12)
Nausea (Gastrointestinal disorders) | 12 (12)
Vomiting (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Constipation (Gastrointestinal disorders) | 6 (6)
Oral mucositis (Gastrointestinal disorders) | 6 (6)
Rash, maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) — Myalgia/arthralgia
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Petechia (Blood and lymphatic system disorders) | 4 (4)
Confusion (Nervous system disorders) | 6 (6)
Hearing impairment (Ear and labyrinth disorders) | 5 (5)
Hypophosphatemia (Investigations) | 1 (1)
alopecia (General disorders) | 11/11 (11)
Anterior uveitis (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only twelve patients were treated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT02379195/Prot_SAP_000.pdf